CLINICAL TRIAL: NCT01225926
Title: A Randomized, Prospective, Multi-Center, Patient-Masked, Bilateral Comparison of Aspheric Toric Intraocular Lens (IOL) Implantation Versus Aspheric Non-Toric Lens Implantation
Brief Title: A Comparison of Aspheric Toric Intraocular Lens (IOL) Implantation Versus Aspheric Non-Toric Lens Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M10-003
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Results first posted 2013-09-24 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Cataract
Keywords: Intraocular Lens; Toric
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toric T3 - T9 (Experimental): AcrySof IQ Toric IOL surgically implanted in the capsular bag of the eye following cataract removal. Both eyes were implanted, with the second eye implanted at least 1 week after and within 1 month of the first eye.
  Interventions: Device: Toric T3 - T9
- IQ SN60WF (Active Comparator): AcrySof IQ IOL surgically implanted in the capsular bag of the eye following cataract removal. Both eyes were implanted, with the second eye implanted at least 1 week after and within 1 month of the first eye.
  Interventions: Device: IQ SN60WF

INTERVENTIONS:
Device: Toric T3 - T9 — Commercially available, acrylic, multifocal IOL intended to provide visual correction over the lifetime of the cataract patient
  Other Names: AcrySof® IQ Toric IOL Models SN6AT3, SN6AT4, SN6AT5, SN6AT6, SN6AT7, SN6AT8, or SN6AT9
  Arms: Toric T3 - T9
Device: IQ SN60WF — Commercially available, acrylic, monofocal IOL intended to provide visual correction over the lifetime of the cataract patient
  Other Names: AcrySof® IQ IOL Model SN60WF
  Arms: IQ SN60WF

SUMMARY:
The purpose of this study was to evaluate and compare uncorrected distance visual acuity measurement in pseudophakic subjects with bilateral implantation of an AcrySof IQ Toric Intraocular Lens (IOL) versus bilateral implantation of an AcrySof IQ IOL.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign an informed consent;
* Willing and able to attend post-operative examinations per protocol schedule;
* In good ocular health, with the exception of cataracts;
* Age-related cataracts in both eyes that require extraction followed by implantation of an intraocular lens;
* Pre-operative corneal cylinder of greater than or equal to 0.75 diopter as determined by auto keratometry;
* In good ocular health, with the exception of cataracts;
* Free of diseases/conditions listed in the precautions of the AcrySof® Toric and AcrySof® IQ package inserts;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Previous corneal surgery;
* Corneal abnormality that would prevent stable and reliable visual acuity and refractive measures;
* Planned multiple procedures during cataract/IOL implantation surgery;
* Ocular disease and/or condition that may compromise study results;
* Ocular trauma, infections or nasolacrimal drainage system malfunction within 3 months of enrolment;
* Pregnant or planning pregnancy during course of study;
* Participation in any other investigational study within 30 days prior to enrolment;
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one study center located in Russia.
Period: Overall Study
Arm/Group | Toric T3 - T9 | IQ SN60WF
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toric T3 - T9 | IQ SN60WF | Total
Number analyzed (Participants) | 12 | 12 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 48.2 (18.64) | 55.5 (16.52) | 51.8 (17.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Monocular Uncorrected Distance Visual Acuity (Monocular UCDVA) at Month 3
Description: Uncorrected visual acuity (i.e., visual acuity measured without spectacles or other visual corrective devices) was assessed using Early Treatment Diabetic Retinopathy Study charts at 100% contrast and measured in logarithm of the minimum angle of resolution (logMAR). Each eye was assessed, and both eyes contributed to the mean. LogMAR 0.00 is equivalent of 20/20 and LogMAR 1.0 is equivalent of 20/200. A more negative logMAR value would indicate a greater improvement in visual acuity.
Time Frame: Month 3
Population: Per protocol: All subjects who received IOLs in both eyes and followed the protocol with no major protocol deviations.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Toric T3 - T9 | IQ SN60WF
Number analyzed (Participants) | 11 | 12
logMAR | 0.089 (0.1212) | 0.225 (0.1503)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. An adverse event was defined as any untoward medical occurrence in a subject regardless of whether or not the event had a causal relationship with the medical device under investigation.
Description: The safety population included all enrolled subjects who received at least one IOL and reported at least one safety assessment.
Arm/Group | Toric T3 - T9 | IQ SN60WF
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toric T3 - T9 (N=12) | IQ SN60WF (N=12)
IOL shift on 10-15 degrees (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was considered a pilot study and did not have an expectation to meet any of the study endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.